CLINICAL TRIAL: NCT01327040
Title: Sensitization of Human Circadian Responses to Light
Brief Title: Light Sensitization Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeanne Duffy, Associate Neuroscientist, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2010-P-000346; R01HL094654 (NIH)
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Chronobiology Disorders; Circadian Rhythm Disorders; Sleep Disorders, Circadian Rhythm
Keywords: light; melatonin; circadian; delayed sleep phase disorder; circadian light sensitivity; circadian timing system
MeSH Terms: conditions — Chronobiology Disorders; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- sensitization duration 1.375h (Experimental): This group will experience a 1.375h sensitization duration prior to the 12h light exposure
  Interventions: Other: light exposure
- sensitization duration 5.5h (Experimental): This group will experience a 5.5h sensitization duration prior to the 12h light exposure
  Interventions: Other: light exposure
- sensitization duration 22h (Experimental): This group will experience a 22h sensitization duration prior to the 12h light exposure
  Interventions: Other: light exposure
- sensitization duration 0.33h (Experimental): This group will experience a 0.33h sensitization duration prior to the 12h light exposure
  Interventions: Other: light exposure

INTERVENTIONS:
Other: light exposure — 12-hour light exposure of approximately 200 lux

SUMMARY:
Circadian rhythm disorders are a class of sleep disorders characterized by misalignment between the timing of sleep and the timing of rhythms driven by the biological clock. Light therapy can effectively treat these disorders, but the intensity and duration of light exposure required to do so has limited its practical use. In this study the investigators will test whether pre-exposure to dim light may enhance the response of the circadian system to light therapy. If so, this could result in shorter treatments that would have greater practical applications.

DETAILED DESCRIPTION:
Sleep disorders affect 35-40% of adults, resulting in diminished quality of life, and increased morbidity, mortality, and risk of automobile and occupational accidents. Circadian rhythm sleep disorders form a distinct class of sleep disorders characterized by misalignment between the timing of sleep and the circadian pacemaker. While light therapy can be an effective treatment of circadian rhythm sleep disorders, there are numerous practical limitations.

Light is the most powerful signal from the environment that influences and regulates daily biological rhythms. It is well-established that the irradiance, duration, and timing of light exposure all affect the response of the circadian system. While it was once thought that these responses were mediated through the visual system, it is now known that there is a network of intrinsically photosensitive retinal ganglion cells (ipRGCs) that mediate circadian responses to light. Other new studies have demonstrated that recent light exposure history affects the circadian response to light in humans.

These recent findings have important implications for the use of light to treat circadian rhythm disorders, including delayed and advanced sleep phase disorders, shift work sleep disorder, and jet lag, and they may also have relevance for the use of light to treat seasonal affective disorder. Up to now, little attention has been paid to the duration or intensity of light exposure prior to such light treatments. The investigators now have evidence that the human circadian system can become desensitized to light during long exposures and evidence that it can be sensitized to light by prior exposure to dim light. These recent findings suggest that light treatment protocols that sensitize the circadian system prior to the light treatment will be more effective than those currently in use.

The 13-day inpatient studies the investigators propose will examine the effect on the human circadian system of different durations of dim-light sensitization prior to a standardized light treatment. These results will be compared within subjects in a randomized cross-over design study in which each subject will receive a control treatment and a light treatment with prior dim-light sensitization. The investigators will also include circadian phase disorder patients to test these mechanisms in the target patient population. Our findings will provide an important step in understanding how new knowledge about the circadian photoreceptive system can be used to refine and provide better treatment options for circadian rhythm disorders.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults with conventional and regular sleep-wake timing
* non-smokers
* completion of medical, psychological, ophthalmological, and sleep screening tests
* able to spend 13 consecutive days/nights in the laboratory

Exclusion Criteria:

* history of neurological or psychiatric disorder
* history of eye injury, eye surgery, or visual disorder (corrective lenses are acceptable)
* history of sleep disorder or regular use of sleep-promoting medication
* current prescription, herbal, or over-the-counter medication use (oral contraceptives are acceptable)

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-10; Primary Completion 2015-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
circadian phase timing | During inpatient study, on days 6-7 and 11-12
  timing of circadian phase as assessed using melatonin and temperature data

SECONDARY OUTCOMES:
melatonin suppression | During inpatient study, on days 6-7 and 11-12
  percent of melatonin suppression

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Czeisler, PhD, MD, Principal Investigator — Brigham and Women's Hospital; Jeanne F Duffy, PhD, Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No